CLINICAL TRIAL: NCT02666690
Title: Study of the Intra-patient Variability of the Quantitative Parameters of Tumor Perfusion Evaluated With Ultrasound Contrast
Acronym: VARIA-DCE-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2010-A01527-32; 2010/1703 (Other: CSET number)
Record Dates: First submitted 2015-08-03; First posted 2016-01-28 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: GIST Metastatic Cancer; Breast Metastatic Cancer; Kidney Metastatic Cancer; Colon Metastatic Cancer; Rectal Metastatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with metastatic cancer treated with anti angiogenics (Experimental)
  Interventions: Device: CEUS (Contrast-enhanced ultrasound)

INTERVENTIONS:
Device: CEUS (Contrast-enhanced ultrasound) — Each patient will be performed 2 contrast echocardiography (a pre-prandial - a post-prandial) before the antiangiogenic treatment, at D15 and D30.

SUMMARY:
RECIST criteria for evaluating tumor response are often inadequate for the evaluation of anti-angiogenic drugs. An evaluation model of tumor perfusion with contrast-enhanced ultrasonography was developed at Gustave Roussy. It assesses the tumor vascular response through the analysis of 7 different parameters. Several studies (four at IGR, involving 117 patients, and a multicenter study involving 400 patients) showed that CEUS allows early evaluation of the effect of anti-angiogenic drugs. Two of these parameters are particularly interesting for the early identification of patients responding (or not) to treatment. Those are area under curve , and area under the wash-out. To further validate the use of these parameters, it is essential to measure and describe the level of their intra-patient variability.

ELIGIBILITY:
Inclusion Criteria:

1. Patient being treated at IGR for metastatic cancer by anti-angiogenic (s) drug (s) in the following indications:

   * Gastrointestinal sarcoma (GIST)
   * Breast Cancers
   * Kidney Cancers
   * Colorectal Cancers
   * Melanoma

   These anti-angiogenic drugs are used alone or in combination: Bevacizumab (Avastin), imatinib (Gleevec), Sorafenib (Nexavar), sunitinib (Sutent), Everolimus (Afinitor) Temsirolimus (Torisel), ... (non exhaustive list).
2. With at least one clearly identified metastatic tumor lesion (and accessible to ultrasound for acquisition 3 minutes without losing the target), measuring more than 2 cm, less than 50% of the volume is necrotic.

   Metastatic lesions are:
   * Liver (30 patients)
   * Or outside the liver (30 patients)
3. Physiological Age: 18-80 years
4. performance status <2
5. Patient information and signature of informed consent

Exclusion Criteria:

1. Background known hypersensitivity to sulfur hexafluoride or one of the components,
2. recent history of acute coronary syndrome or unstable ischemic heart disease,
3. Acute heart failure, heart failure stage III or IV, or severe rhythm disorders,
4. uncontrolled hypertension or severe pulmonary hypertension,
5. Right-Left Shunt,
6. Respiratory Distress Syndrome,
7. Patient without vascularized tumor (without contrast enhancement)
8. patient whose antiangiogenic has already started,
9. Pregnant woman likely to be or breastfeeding,
10. Persons deprived of liberty or under guardianship,
11. Unable to submit to medical monitoring of the trial for geographical, social or psychological reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Variability of quantitative parameters of Tumor Perfusion Evaluated With Ultrasound Contrast | Assessed 30 days after inclusion
  Demonstrate that for the hepatic metastatic sites and for non hepatic metastatic sites the variability of the measured quantitative parameters on two different perfusion curves is less than 30%

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France